CLINICAL TRIAL: NCT03920176
Title: Computed Tomography Coronary Angiography for the Prevention of Myocardial Infarction (The SCOT-HEART 2 Trial)
Acronym: SCOT-HEART 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRAS ID: 261185
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiology; Computed tomography coronary angiography
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computed tomography coronary angiography (Active Comparator)
  Interventions: Diagnostic Test: Computed tomography coronary angiography
- Assign Score only (Sham Comparator)
  Interventions: Other: ASSIGN Score

INTERVENTIONS:
Diagnostic Test: Computed tomography coronary angiography — CTCA >64 detector row scanner
  Arms: Computed tomography coronary angiography
Other: ASSIGN Score — ASSIGN Cardiovascular Risk Score
  Arms: Assign Score only

SUMMARY:
It is hypothesised that, in individuals being considered for cardiovascular preventative therapy, computed tomography coronary angiography guided management will reduce the future risk of coronary heart disease death or non-fatal myocardial infarction compared to management guided by the current standard of care, a cardiovascular risk score.

DETAILED DESCRIPTION:
Prevention of cardiovascular disease is currently guided by probabilistic risk scores that both over and under treat individuals, commit most middle-aged people to pharmacotherapy, and have little evidence base. It has been demonstrated that use of computed tomography coronary angiography (CTCA) is associated with changes in the diagnosis and treatment of patients presenting with stable chest pain, and that this leads to a marked reduction in the future risk of myocardial infarction. Importantly, the proportionate reduction in coronary events was most marked in those with non-anginal chest pain irrespective of their cardiovascular risk score which again demonstrated poor discrimination. The research team propose a randomised controlled trial of at least 6,000 middle-aged individuals at risk of cardiovascular disease that will compare these two strategies of targeting preventative therapies: a probabilistic cardiovascular risk score, and screening with CTCA. This trial will determine if CTCA guided management will be associated with better targeted intervention, prevent over medicating the general population, and result in fewer future coronary heart disease events than the current standard of care using a cardiovascular risk score.

ELIGIBILITY:
INCLUSION CRITERIA

* ≥40 and ≤70 years of age
* Resident in Scotland and have a Community Health Index (CHI) number
* One or more of the following risk factors:

  * >60 years of age
  * Current or recent (within 12 months) smoker
  * Clinical diagnosis of hypertension
  * Known hypercholesterolaemia or total cholesterol >6.0 mmol/L or receiving statin therapy
  * Diabetes mellitus
  * Rheumatoid arthritis
  * Systemic lupus erythematosus (SLE)
  * Family history of premature cardiovascular disease (first degree relative with atherosclerotic cardiovascular disease below 60 years)
  * Chronic kidney disease stage 3 (estimate glomerular filtration rate 30-59 mL/min/1.73 m2).

EXCLUSION CRITERIA

* Inability to undergo CTCA
* Known coronary heart disease or other major atherosclerotic cardiovascular disease
* Prior invasive or non-invasive coronary angiography within the last 5 years
* Chronic kidney disease stage ≥4 (estimate glomerular filtration rate <30 mL/min/1.73 m2)
* Known homozygous familial hypercholesterolaemia or other serious inherited disorders of lipid metabolism requiring statin therapy
* Intolerance of all statins
* Statin therapy for >2 years.
* Previous coronary artery imaging completed specifically for cardiovascular risk assessment with a result of >10 AU.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6139 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary heart disease death or non-fatal myocardial infarction | 5 years
  The primary research objective of the trial is to determine whether, in individuals with risk for cardiovascular disease, coronary heart disease screening with CTCA is associated with a reduction in the rate of coronary heart disease death or non-fatal myocardial infarction when compared to a probabilistic cardiovascular risk score approach.

SECONDARY OUTCOMES:
Death | 5 Years
  Number of all-cause, cardiovascular, coronary heart disease and non-cardiovascular deaths
Cardiovascular Events | 5 Years
  Number of participants who have fatal and non-fatal myocardial infarction or stroke
Cardiovascular Procedures | 5 Years
  Number of Invasive coronary angiography and coronary revascularisation procedures
Quality of Life (EQ-5D-5L) | 2 Years
  Quality of life measured using EQ-5D-5L instrument
Prescription | 5 Years
  Rates of prescription of preventative therapies (anti-platelet, statin and angiotensin-converting enzyme inhibitor therapies)
Lifestyle Modification | 2 Years
  Uptake of lifestyle modifications (smoking, exercise and diet) measured using self-reported questionnaire
Health Economics | 2 Years
  Health economic assessment of cost-effectiveness
Cholesterol | 5 Years
  Serum cholesterol concentration
Disadvantages of CTCA- Radiation | 5 Years
  Radiation dose (mGy-cm)
Disadvantages of CTCA- incidental findings | 5 Years
  Number of participants with incidental findings from CTCA

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, Principal Investigator — University of Edinburgh
Locations (1):
- Western General Hospital, Edinburgh, City Of Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The intention is to share anonymised data with external collaborators and scientists. The data will be available one year after the primary paper has been published (anticipated to be in 2027) .
Supporting Information: Study Protocol, CSR
Time Frame: After 2027.
Access Criteria: Requests can be made by email from 2027.

REFERENCES:
- See also: Study website — https://www.ed.ac.uk/usher/edinburgh-clinical-trials/our-studies/ukcrc-studies/scot-heart-2

DOCUMENTS (1):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03920176/Prot_001.pdf